CLINICAL TRIAL: NCT01234402
Title: An Open-Label, Multicenter, Randomized Phase 2 Study Evaluating the Safety and Efficacy of Ramucirumab (IMC-1121B) Drug Product or Icrucumab (IMC-18F1) in Combination With Capecitabine or Capecitabine Monotherapy, in Unresectable, Locally Advanced or Metastatic Breast Cancer Patients Previously Treated With Anthracycline and Taxane Therapy
Brief Title: Study of Icrucumab (IMC-18F1) or Ramucirumab Drug Product (DP) in Combination With Capecitabine or Capecitabine on Previously Treated Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13944; CP20-0903 (Other: ImClone LLC); I4Y-IE-JCDD (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ramucirumab; IMC-18F1; Icrucumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ramucirumab DP + Capecitabine (Experimental): Cycles repeat until disease progression, the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant.
  Interventions: Biological: Ramucirumab DP; Drug: Capecitabine
- Icrucumab + Capecitabine (Experimental): Cycles repeat until disease progression, the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant.
  Interventions: Biological: IMC-18F1; Drug: Capecitabine
- Capecitabine* (Active Comparator): Crossover Study:
  * At the discretion of the investigator, participants will be eligible to receive either ramucirumab DP or Icrucumab (IMC-18F1) in combination with capecitabine, after radiographic disease progression while on capecitabine. The investigator will decide which investigational product will be given.
  Cycles repeat every 21 days until disease progression, the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Biological: Ramucirumab DP — 10 mg/kg I.V.
  Day 1 of every-21-day cycle
  Other Names: IMC-1121B; LY3009806
  Arms: Ramucirumab DP + Capecitabine
Biological: IMC-18F1 — 12 mg/kg I.V.
  Days 1 and 8 of every-21-day cycle
  Other Names: Icrucumab; LY3012212
  Arms: Icrucumab + Capecitabine
Drug: Capecitabine — 1000 mg/m^2 orally
  Twice a day for 14 days

SUMMARY:
An open-label, multicenter, randomized, Phase 2 trial in which participant with unresectable, locally advanced or metastatic breast cancer who have been previously treated with anthracycline and taxane therapy receive ramucirumab DP or Icrucumab (IMC-18F1) administered on an every-21-day cycle (in combination with oral capecitabine therapy; capecitabine is administered twice a day on Days 1-14 of each cycle). Approximately 150 participants will be randomized in a 1:1:1 ratio to either ramucirumab DP or Icrucumab (IMC-18F1) in combination with capecitabine (Arm A and Arm B, respectively) or capecitabine monotherapy (Arm C). Randomization will be stratified by triple-negative receptor status (estrogen receptor-negative, progesterone receptor-negative, and human epidermal growth factor receptor-2 [HER2/neu]-negative) (yes/no) and receipt of prior antiangiogenic therapy.

Treatment with the study medication(s) will continue until disease progression, the development of unacceptable toxicity, noncompliance or withdrawal of consent by the participant, or investigator decision. Capecitabine dose reductions in the setting of significant myelosuppression, hand-and-foot syndrome, or diarrhea will be required.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed breast cancer which at the time of study entry is either Stage III disease not amenable to curative therapy or Stage IV disease
* Has measurable or nonmeasurable disease
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Has received prior anthracycline therapy
* Has received prior taxane therapy
* Participants with human epidermal growth factor receptor-2 (HER2) positive disease must have progressed on or following trastuzumab
* Participants with hormone receptor-positive disease must have progressed on or following hormone therapy
* Has received ≤ 3 prior chemotherapy regimens in any setting (a regimen is defined as any agent[s] that has been administered for more than 1 cycle; sequential neoadjuvant/adjuvant treatment is considered 1 regimen)
* Has completed any prior radiotherapy ≥ 4 weeks prior to randomization
* Has completed any prior hormonal therapy ≥ 2 weeks prior to randomization
* Has adverse events (AEs) that have resolved to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v 4.0) from all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy,or hormonal therapy
* Has adequate hematologic, coagulation, hepatic and renal function
* Does not have:

  * cirrhosis at a level of Child-Pugh B (or worse) or
  * cirrhosis (any degree) and a history of hepatic encephalopathy or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis
* Has urinary protein is ≤ 1+ on dipstick or routine urinalysis; if urine protein ≥ 2+, a 24-hour urine collection must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study
* Agrees to use adequate contraception during the study period and for 12 weeks after the last dose of study medication

Exclusion Criteria:

* Has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer, curatively treated cervical carcinoma in situ, or other noninvasive carcinoma or in situ neoplasm. A participant with previous history of malignancy is eligible, provided that there has been a disease-free interval for > 3 years
* Has a known sensitivity to capecitabine, any of its components, or other drugs formulated with polysorbate 80
* Has a known sensitivity to 5-fluorouracil (5-FU)
* Has a known dihydropyrimidine dehydrogenase deficiency
* Has received prior capecitabine treatment for advanced breast cancer
* Has received investigational therapy within 2 weeks prior to randomization
* Has received bevacizumab within 4 weeks prior to randomization
* Has received more than 1 prior antiangiogenic agent for breast cancer
* Has a known sensitivity to agents of similar biologic composition as ramucirumab DP or Icrucumab (IMC-18F1), or other agents that specifically target vascular endothelial growth factor (VEGF)
* Has an acute/subacute bowel obstruction or history of chronic diarrhea requiring ongoing medical intervention
* Has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
* Has experienced a Grade ≥ 3 bleeding event within 3 months prior to randomization
* Is receiving prophylactic or therapeutic anticoagulation with warfarin or any other oral anticoagulant
* Has an uncontrolled intercurrent illness, including, but not limited to uncontrolled hypertension, symptomatic anemia, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorder in the opinion of the investigator
* Has experienced any arterial thrombotic or thromboembolic events, including, but not limited to myocardial infarction, transient ischemic attack, or cerebrovascular accident within 6 months prior to randomization
* Has brain metastases, uncontrolled spinal cord compression, or leptomeningeal disease
* Has an ongoing or active infection requiring parenteral antibiotic, antifungal, or antiviral therapy
* Has received a prior allogeneic organ or tissue transplantation
* Has undergone major surgery within 4 weeks prior to randomization, or subcutaneous venous access device placement within 7 days prior to randomization
* Has had a serious nonhealing wound, ulcer, or bone fracture within 4 weeks prior to randomization
* Has known HIV or AIDS infection
* Has an elective or planned major surgery to be performed during the course of the trial
* Participant is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2011-03; Primary Completion 2013-10 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- United States (20):
  - ImClone Investigational Site, Scottsdale, Arizona
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Augusta, Georgia
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Baton Rouge, Louisiana
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Stony Brook, New York
  - ImClone Investigational Site, The Bronx, New York
  - ImClone Investigational Site, Washington, North Carolina
  - ImClone Investigational Site, Cincinnati, Ohio
  - ImClone Investigational Site, Columbus, Ohio
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, San Antonio, Texas
  - ImClone Investigational Site, Salt Lake City, Utah
  - ImClone Investigational Site, Richmond, Virginia
  - ImClone Investigational Site, Spokane, Washington
  - ImClone Investigational Site, Morgantown, West Virginia
- Canada (3):
  - ImClone Investigational Site, Calgary, Alberta
  - ImClone Investigational Site, Edmonton, Alberta
  - ImClone Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Vahdat LT, Layman R, Yardley DA, Gradishar W, Salkeni MA, Joy AA, Garcia AA, Ward P, Khatcheressian J, Sparano J, Rodriguez G, Tang S, Gao L, Dalal RP, Kauh J, Miller K. Randomized Phase II Study of Ramucirumab or Icrucumab in Combination with Capecitabine in Patients with Previously Treated Locally Advanced or Metastatic Breast Cancer. Oncologist. 2017 Mar;22(3):245-254. doi: 10.1634/theoncologist.2016-0265. Epub 2017 Feb 20. PMID 28220020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in Capecitabine arm were allowed to cross-over to ramucirumab or icrucumab in combination with capecitabine, after radiographic disease progression while on capecitabine.
Pre-assignment Details: Completers are those participants who died or alive and on study at conclusion but off treatment.
Groups:
- Ramucirumab + Capecitabine: Participants received 10 milligram per kilogram (mg/kg) Ramucirumab intravenously on day 1 of 21 days cycle along with 1000 milligram per square meter (mg/m^2) of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
- Icrucumab + Capecitabine: Participants received 12 mg/kg Icrucumab intravenously on day 1 and day 8 of 21 day cycle along with 1000 mg/m^2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
- Capecitabine: Participants received 1000 mg/m^2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
  After radiographic diseases progression while on Capecitabine, participants were crossed-over to either Ramucirumab or Icrucumab;
  Participants crossed-over to Ramucirumab + Capecitabine had received 10 mg/kg Ramucirumab intravenously on day 1 of 21 days cycle along with 1000 mg/m^2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
  Participants crossed-over to Icrucumab + Capecitabine received 12 mg/kg Icrucumab intravenously on day 1 and day 8 of 21 day cycle along with 1000 mg/m^2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
Period: Overall Study
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Started | 52 | 51 | 50
Received at Least One Dose of Study Drug | 52 | 49 | 49
Capecitabine Crossover to Ramucirumab | 0 | 0 | 29
Capecitabine Crossover to Icrucumab | 0 | 0 | 1
Completed | 51 | 45 | 42
Not Completed | 1 | 6 | 8
Not completed — Lost to Follow-up | 0 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3 | 4
Not completed — Never treated: Death | 0 | 0 | 1
Not completed — Never treated: Withdrawal By Subject | 0 | 1 | 0
Not completed — Never treated: Insurance Denied Xeloda | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Ramucirumab + Capecitabine: Participants received 10 mg/kg Ramucirumab intravenously on day 1 of 21 days cycle along with 1000 mg/m^2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
- Total: Total of all reporting groups
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine | Total
Number analyzed (Participants) | 52 | 49 | 49 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (10.75) | 51.1 (11.54) | 53.5 (11.12) | 53.3 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 49 | 149
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 6
  Not Hispanic or Latino | 49 | 44 | 45 | 138
  Unknown or Not Reported | 1 | 2 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  American Indian or Alaska Native,White | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 1 | 4
  Black or African American | 13 | 8 | 4 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  White | 36 | 37 | 39 | 112
  White, Other | 0 | 0 | 1 | 1
  Other | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until the date of objectively determined progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death from any cause, whichever is first. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 millimeter (mm) and the appearance of ≥1 new lesions was progression. Participants who did not progress, were lost to follow-up, or had missed 2 or more scheduled tumor assessments were censored at the day of their last adequate tumor assessment.
Time Frame: From Date of Randomization until Disease Progression or Death Due to Any Cause (Up To 97 weeks)
Population: All randomized participants who received at least one dose of study drug; Censored participants: Ramucirumab + Capecitabine = 12; Icrucumab + Capecitabine = 11; Capecitabine = 7
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 52 | 49 | 49
Weeks | 22.1 [12.1 to 36.1] | 7.3 [6.3 to 13.0] | 19.0 [12.1 to 24.3]
Statistical Analysis 1: Comparison: Ramucirumab + Capecitabine vs Capecitabine; Kaplan-Meier methodology estimated median PFS; Test type: Other; p = 0.1315, Log Rank; Hazard Ratio (HR) = 0.691, 95% CI 2-sided [0.429 to 1.114]
Statistical Analysis 2: Comparison: Icrucumab + Capecitabine vs Capecitabine; Kaplan-Meier methodology estimated median PFS; Test type: Other; p = 0.0851, Log Rank; Hazard Ratio (HR) = 1.480, 95% CI 2-sided [0.938 to 2.335]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death from any cause. If the participant is alive at the end of the follow-up period or is lost to follow-up, OS will be censored on the last date the participant is known to be alive.
Time Frame: From Date of Randomization until Death Due to Any Cause (Up To 160 weeks)
Population: All randomized participants who received at least one dose of study drug; censored participants: Ramucirumab + Capecitabine = 21; Icrucumab + Capecitabine = 17; Capecitabine = 22 Participants were analyzed as per the randomization.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 52 | 49 | 49
Weeks | 67.4 [41.3 to 82.6] | 62.1 [41.0 to 84.0] | 71.6 [57.4 to 89.7]
Statistical Analysis 1: Comparison: Ramucirumab + Capecitabine vs Capecitabine; Test type: Other; p = 0.0283, Log Rank; Hazard Ratio (HR) = 1.833, 95% CI 2-sided [1.060 to 3.169]
Statistical Analysis 2: Comparison: Icrucumab + Capecitabine vs Capecitabine; Test type: Other; p = 0.1550, Log Rank; Hazard Ratio (HR) = 1.468, 95% CI 2-sided [0.862 to 2.501]

3. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: The ORR is the number of all participants with Partial Response (PR) or Complete Response (CR) according to RECIST v1.1 from the start of the treatment until disease progression/recurrence. CR was defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm. PR was defined as ≥30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, taking as reference smallest sum on study (included baseline sum if that was the smallest on study); sum must have demonstrated an absolute increase of ≥5 mm and the appearance of ≥1 new lesions was progression.
Time Frame: From Date of Randomization until Disease Progression/Recurrence (Up to 97 weeks)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 52 | 49 | 49
Percentage of Participants | 28.8 [17.1 to 43.1] | 20.4 [10.2 to 34.3] | 34.7 [21.7 to 49.6]
Statistical Analysis 1: Comparison: Ramucirumab + Capecitabine vs Capecitabine; Test type: Other; p = 0.6691, Fisher Exact
Statistical Analysis 2: Comparison: Icrucumab + Capecitabine vs Capecitabine; Test type: Other; p = 0.1743, Fisher Exact

4. Secondary Outcome: Duration of Response
Description: Duration of response is measured from the time measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that the criteria for progressive disease (PD) is met (taking as a reference for PD that smallest measurement recorded since the treatment started), or death, is objectively documented.CR was defined as the disappearance of all non-nodal target lesions, with the short axes of any target lymph nodes reduced to <10 mm. PR was defined as ≥30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph nodes), taking as reference the baseline sum diameter.PD defined as ≥20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Sum must also have demonstrated an absolute increase of ≥5 mm, or the appearance of 1 or more new lesions was considered progression.
Time Frame: From Date of CR, PR until Disease Progression or Death Due to Any Cause (Up To 97 weeks)
Population: All randomized participants who received at least one dose of study drug and had CR/PR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 15 | 10 | 17
weeks | 43.1 [12.0 to 49.0] | 20.1 [1.9 to 33.9] | 17.1 [6.4 to 30.7]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse event (AE) will be regarded as treatment-emergent if onset date occurs any time on or after the administration of the first dose of study treatment up to 30 days after the last dose of study treatment (or up to any time if related to study treatment); or it occurs prior to first dose date and worsens while on therapy or up to 30 days after the last dose of study treatment (or up to any time if related to study treatment).
  A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Up To 160 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 52 | 49 | 49
Participants | 52 | 49 | 48

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE was defined as any untoward medical occurrence that at any dose:
  Resulted in death; Was life-threatening; Required inpatient hospitalization or caused prolongation of existing hospitalization; Resulted in persistent or significant disability/incapacity; Was a congenital anomaly/birth defect; Required intervention to prevent permanent impairment/damage; Was an important medical event (defined as a medical event that may not have been immediately life-threatening or resulted in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention to prevent one of the other serious outcomes listed in the definition above).
  A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Up To 160 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine
Number analyzed (Participants) | 52 | 49 | 49
Participants | 20 | 25 | 6

7. Secondary Outcome: Maximum Concentration (Cmax) Ramucirumab Drug Product (DP) or Icrucumab
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: For ramucirumab, all randomized participants who received at least one dose of study drug & had evaluable pharmacokinetic (PK) samples.
  For icrucumab, zero participants analyzed as reliable PK parameters could not be estimated using non-compartmental PK analysis due to insufficient number of samples.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 11 | 0
Microgram per milliliter | 308 (25) |

8. Secondary Outcome: Minimum Concentration (Cmin) Ramucirumab Drug Product (DP) or Icrucumab
Description: Minimum Concentration (Cmin) Ramucirumab Drug Product (DP) or Icrucumab.
Time Frame: Cycle 2,4,6,8,0,12,14,16,18,22: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micro gram per milliliter
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 12 | 0
Micro gram per milliliter
  Cycle 2 | 23.7 (58) |
  Cycle 4: number analyzed (Participants) | 4 | 0
  Cycle 4 | 80.6 (67) |
  Cycle 6: number analyzed (Participants) | 4 | 0
  Cycle 6 | 44.7 (83) |
  Cycle 8: number analyzed (Participants) | 3 | 0
  Cycle 8 | 65.8 (43) |
  Cycle 10: number analyzed (Participants) | 4 | 0
  Cycle 10 | 66.8 (37) |
  Cycle 12: number analyzed (Participants) | 3 | 0
  Cycle 12 | 74.3 (38) |
  Cycle 14: number analyzed (Participants) | 1 | 0
  Cycle 14 | 62.5 |
  Cycle 16: number analyzed (Participants) | 1 | 0
  Cycle 16 | 50.5 |
  Cycle 18: number analyzed (Participants) | 1 | 0
  Cycle 18 | 50.5 |
  Cycle 22: number analyzed (Participants) | 1 | 0
  Cycle 22 | 55.0 |

9. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Infinity of Ramucirumab or Icrucumab
Description: Area Under the Concentration (AUC) Versus Time Curve From Time Zero to Infinity of Ramucirumab and Icrucumab.
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/mL
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 7 | 0
microgram*hour/mL | 54400 (42) |

10. Secondary Outcome: Terminal Half-life (t½) of Ramucirumab or Icrucumab
Description: Terminal half-life (t½) of Ramucirumab and Icrucumab.
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: as for outcome 7
Measure: Geometric Mean (Full Range); unit: Days
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 7 | 0
Days | 6.80 [5.22 to 8.57] |

11. Secondary Outcome: Clearance (Cl) of Ramucirumab or Icrucumab
Description: Clearance (Cl) of Ramucirumab and Icrucumab.
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 7 | 0
Liters per hour | 0.0141 (34) |

12. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ramucirumab or Icrucumab
Description: Volume of Distribution at Steady State (Vss) of Ramucirumab and Icrucumab.
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 11 | 0
Liters | 3.17 (18) |

13. Secondary Outcome: Number of Participants With Anti-Ramucirumab and Anti-Icrucumab Antibodies
Time Frame: Cycle 1: Pre-infusion, 1h, 48h, 72h, 168, 336h post infusion
Population: For ramucirumab, Aall randomized participants who received at least one dose of study drug and had evaluable serum samples for antibody assessment.
  For icrucumab, zero participants analyzed as antibody assessment data was not collected for Icrucumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine
Number analyzed (Participants) | 43 | 0
Participants
  Treatment emergent antibody | 0 |
  Neutralizing antibody | 0 |

ADVERSE EVENTS:
Time Frame: Up To 160 Weeks
Description: All randomized participants who received at least one dose of study drug.
Groups:
- Ramucirumab + Capecitabine; Crossover to Ramucirumab DP + Capecitabine: Participants received 10 milligram per kilogram (mg/kg) Ramucirumab intravenously on day 1 of 21 days cycle along with 1000 milligram per meter square (mg/m*2) of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
- Icrucumab + Capecitabine; Crossover to Icrucumab + Capecitabine: Participants received 12 mg/kg Icrucumab intravenously on day 1 and day 8 of 21 day cycle along with 1000 milligram per meter square (mg/m*2) of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
- Capecitabine: Participants received 1000 mg/m*2 of Capecitabine twice daily orally on days 1 to 14 of 21 days cycle.
Arm/Group | Ramucirumab + Capecitabine | Icrucumab + Capecitabine | Capecitabine | Crossover to Ramucirumab DP + Capecitabine | Crossover to Icrucumab + Capecitabine
Serious Adverse Events (participants affected / at risk) | 20/52 | 25/49 | 6/49 | 5/29 | 0/1
Other Adverse Events (participants affected / at risk) | 51/52 | 49/49 | 48/49 | 29/29 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Capecitabine (N=52) | Icrucumab + Capecitabine (N=49) | Capecitabine (N=49) | Crossover to Ramucirumab DP + Capecitabine (N=29) | Crossover to Icrucumab + Capecitabine (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab + Capecitabine (N=52) | Icrucumab + Capecitabine (N=49) | Capecitabine (N=49) | Crossover to Ramucirumab DP + Capecitabine (N=29) | Crossover to Icrucumab + Capecitabine (N=1)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 14 (35) | 12 (28) | 3 (5) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 7 (13) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (16) | 1 (15) | 3 (15) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (16) | 6 (10) | 6 (10) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (13) | 1 (2) | 9 (10) | 5 (11) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 4 (4) | 6 (6) | 2 (2) | 1 (2) | 0 (0)
Periorbital oedema (Eye disorders) | 2 (2) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (3) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 6 (10) | 4 (6) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 18 (25) | 14 (16) | 17 (25) | 7 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 22 (47) | 20 (38) | 27 (58) | 5 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 5 (6) | 3 (3) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (47) | 37 (53) | 26 (39) | 8 (16) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 14 (20) | 4 (7) | 7 (12) | 5 (6) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (23) | 25 (31) | 14 (25) | 7 (10) | 0 (0)
Asthenia (General disorders) | 6 (7) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Face oedema (General disorders) | 1 (1) | 9 (12) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 27 (54) | 27 (43) | 26 (36) | 11 (15) | 0 (0)
Influenza like illness (General disorders) | 6 (7) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 8 (14) | 4 (6) | 9 (16) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 13 (21) | 19 (37) | 6 (7) | 5 (8) | 1 (1)
Pain (General disorders) | 5 (8) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 14 (18) | 7 (8) | 4 (6) | 5 (6) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 3 (3) | 2 (3) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 7 (13) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (8) | 3 (3) | 4 (6) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (7) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (12) | 1 (1) | 5 (6) | 3 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (14) | 2 (3) | 7 (7) | 2 (6) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 4 (9) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 4 (4) | 2 (12) | 1 (2) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (6) | 2 (2) | 1 (2) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (9) | 2 (3) | 2 (5) | 1 (2) | 1 (1)
Platelet count decreased (Investigations) | 3 (4) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 4 (4) | 1 (2) | 0 (0)
Weight increased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 17 (26) | 11 (16) | 10 (17) | 6 (9) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 7 (7) | 3 (4) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (15) | 4 (7) | 2 (2) | 3 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (8) | 3 (7) | 1 (1) | 3 (4) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (22) | 6 (9) | 4 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (18) | 7 (10) | 12 (17) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4) | 0 (0) | 3 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (19) | 2 (2) | 8 (13) | 3 (4) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (15) | 6 (8) | 8 (9) | 6 (9) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 0 (0) | 5 (5) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 6 (8) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 4 (5) | 3 (3) | 2 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (3) | 0 (0) | 1 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (29) | 3 (3) | 6 (7) | 3 (6) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (8) | 6 (7) | 3 (3) | 3 (4) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (8) | 6 (6) | 3 (3) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 26 (60) | 9 (11) | 11 (18) | 13 (16) | 1 (1)
Migraine (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 10 (17) | 6 (8) | 4 (5) | 2 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 5 (10) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 7 (8) | 5 (6) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 6 (6) | 6 (6) | 4 (6) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 9 (9) | 12 (14) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (7) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (27) | 10 (11) | 9 (10) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (29) | 16 (19) | 9 (10) | 7 (11) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 0 (0) | 3 (3) | 5 (7) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 2 (2) | 2 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3) | 5 (5) | 2 (2) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 9 (10) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 5 (6) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 7 (9) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 (127) | 15 (38) | 35 (114) | 17 (40) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (5) | 2 (2) | 3 (3) | 3 (5) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (13) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (2) | 0 (0) | 4 (8) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 16 (35) | 1 (1) | 1 (1) | 7 (8) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is for five years after the study conclusion/termination, after five years disclosure restriction on PI is that sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.